CLINICAL TRIAL: NCT02947269
Title: A Randomized Double-blind Placebo Controlled Trial of Prucalopride to Reduce the Duration of Postoperative Ileus in Patients Undergoing Elective Colorectal Surgery
Brief Title: Prucalopride in Postoperative Ileus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, A/Prof Ian Bissett, Professor Ian Bissett, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UOA-prucRCT1
Record Dates: First submitted 2016-10-23; First posted 2016-10-27 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Ileus; Colorectal Surgery; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients will receive an oral capsule containing 2mg Prucalopride 2-3 hours preoperatively. Study medication (2mg oral Prucalopride daily) will continue for 6 days postoperatively or until the patient has achieved the study's primary outcome.
  Interventions: Drug: Prucalopride
- Placebo group (Placebo Comparator): Patients will receive an oral capsule containing a placebo 2-3 hours preoperatively. Study medication (placebo) will continue for 6 days preoperatively or until the patient has achieved the study's primary outcome.
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Prucalopride — Prucalopride 2mg capsule
  Other Names: Resolor; Resotrans
  Arms: Intervention group
Drug: Placebo Oral Capsule — Placebo capsule
  Arms: Placebo group

SUMMARY:
Postoperative ileus (POI) refers to the period of gut dysmotility that occurs after abdominal surgery. Patients with POI are unable to eat, suffer ongoing nausea and vomiting, are unable to open their bowels and have a prolonged hospital stay. Research at ADHB shows that 25% of patients will have a prolonged POI after elective bowel resection, which makes it the most common major complication after colorectal surgery. Clinicians currently lack a definitive medication to prevent or treat POI, which means POI causes patients ongoing morbidity and places a significant drain on healthcare resources. Serotonin plays an important role in gut motility. Evidence suggests that serotonin agonists, such as prucalopride, increase gut transit and may have anti-inflammatory properties. The hypothesis of this study is that Prucalopride given pre-operatively and continued post-operatively in patients having an elective bowel resection will improve gut function recovery after surgery and reduce POI.

The investigators' proposed study is a double-blinded randomised controlled trial of prucalopride compared to an identical placebo tablet, in patients having an elective bowel resection at Auckland City Hospital. Patients will receive a single tablet of Prucalopride or placebo 2-3 hours preoperatively and then daily after operation for a maximum of 6 days. The primary endpoint will be return to bowel function defined by the time to tolerate a solid diet and pass stool. In addition, the investigators plan to assess postoperative gastric emptying rates using the safe and non-invasive carbon breath test method. This will allow the investigators to determine the effects of prucalopride on the stomach, and support its role as a gastric prokinetic.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients from Auckland District Health Board catchment
* Age 18 or older
* Elective and subacute surgery
* Right hemicolectomy, left hemicolectomy, sigmoid colectomy, anterior resection, Hartmann's procedure, subtotal colectomy
* Operation with or without the formation of a colostomy
* Indication for operation: colon cancer, diverticular disease, gynaecological
* Able to understand risks and benefits of the study
* Able to give informed consent

Exclusion Criteria:

* ASA 4 or greater
* Allergy to any serotonin medication
* Active inflammatory bowel disease
* Planned formation of an ileostomy during surgery
* Moderate to severe renal impairment (Creatinine clearance<50mL/min/1.73m2)
* Severe hepatic impairment (Child-Pugh C)
* Pregnancy
* Pre-existing gut dysmotility disorder including endocrine, metabolic or neurological cause
* Pre-operative malnutrition requiring parenteral nutrition
* Inability to give consent or participate in post-operative assessments due to dementia, cognitive impairment, language difficulties, delirium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Time until recovery of gastrointestinal function | From date of surgery until discharge from hospital (14 days on average)
  Recovery of GI function is defined by the later time point (in days) of time to passage of stool AND time to tolerance of a solid or semi-solid diet. Patients will be reviewed twice per day using a structured questionnaire.

SECONDARY OUTCOMES:
Time until passage of stool (in days) | From date of surgery until discharge from hospital (14 days on average)
Time until passage of flatus (in days) | From date of surgery until discharge from hospital (14 days on average)
Time until tolerance of solid oral diet (in days) | From date of surgery until discharge from hospital (14 days on average)
Presence of prolonged postoperative ileus | From date of surgery until discharge from hospital (14 days on average)
  Prolonged postoperative ileus is defined as presence of 2 or more of the following criteria on or after day 4 postoperatively: nausea or vomiting, inability to tolerate a solid or semi-solid oral diet, abdominal distension, absence of flatus and stool, radiological evidence of ileus.
Levels of serum inflammatory markers (in pg/mL) | Inflammatory markers will be collected preoperatively, day 1 and 3 postoperatively. Blood samples will be stored after collection for later testing (up to 1 year).
  Markers to be tested: CRP, IL1beta, IL6, IL8, IL12, TNFalpha
Length of postoperative stay (in days) | From date of surgery until discharge from hospital (14 days on average)

OTHER OUTCOMES:
Rate of gastric emptying using the 13-carbon octanoate breath test | This test will be undertaken on day 2 postoperatively, and will take approximately 4 hours
  A subgroup of 40 patients will be investigated for this study

CONTACTS AND LOCATIONS:
Locations (1):
- University of Auckland, Auckland, New Zealand

REFERENCES:
- [Derived] Milne T, Liu C, O'Grady G, Woodfield J, Bissett I. Effect of prucalopride to improve time to gut function recovery following elective colorectal surgery: randomized clinical trial. Br J Surg. 2022 Jul 15;109(8):704-710. doi: 10.1093/bjs/znac121. PMID 35639621